CLINICAL TRIAL: NCT05480982
Title: Cognitive Functional Therapy Compared With Pilates in Elderly Patients With Chronic Low Back Pain Treated Via Telerehabilitation: A Randomized Controlled Trial
Brief Title: Cognitive Functional Therapy Compared With Pilates in Elderly Patients With Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Universitário Augusto Motta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CFT/PILATES/TELE
Record Dates: First submitted 2022-05-27; First posted 2022-07-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Low Back Pain
Keywords: low back pain; cognitive functional therapy; telehealth; Pilates; behavioral therapy; exercise therapy
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial with allocation of two parallel groups
Who Masked: Investigator
Masking Description: The assessors were not considered blinded because participants were not blinded and outcomes were self-reported. However, to guarantee that the treatment expectation was evenly balanced between the groups and decrease measurement bias, the participants did not know the study hypothesis, and the assessors did not know the participant's intervention group. The statistician was blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive functional therapy (CFT) via tele rehabilitation (Experimental): Cognitive Functional Therapy (CFT) is a physiotherapy-led intervention which has evolved from an integration of foundational behavioral psychology and neuroscience within the physiotherapy practice directed at the multidimensional biopsychosocial nature of low back pain. The clinical journey is adapted to the individual's profile following three main components: (i) making sense of pain, (ii) exposure with control and (iii) lifestyle changes.
  The first 2 one-hour treatment sessions of CFT will be delivered individually and via videoconference in a weekly basis. The following one-hour treatment sessions (from 6 to 9 sessions) will be delivered in groups (up to 6 participants). One group booster session will be delivered 20 weeks after randomization
  Interventions: Behavioral: Cognitive functional therapy via tele rehabilitation
- Pilates (Active Comparator): Participants in the comparison group will receive Pilates method using classic principles and exercises recommended by Joseph Pilates. No specific accessories or equipment will be used, allowing the exercises to be performed under any circumstances. Based on Pilates, 10 exercises were selected: Leg Pull Front, One Leg Circle, One Leg Kick, One leg stretch, Shoulder bridge, Side bend, Spine Stretch , Swimming, The hundred and The Saw. The main objective of the exercises is to improve physical capacities, including mobility, flexibility, muscle strength and activation of the "power house" center of force, with the therapeutic aim of a positive evolution of chronic non-specific low back pain. The one-hour sessions will be delivered once a week. Participants will be instructed to perform the set of exercises once a week without the supervision of the physiotherapist. The number of group sessions (up to 6 participants) will vary between 8 to 12.
  Interventions: Other: Pilates via tele rehabilitation

INTERVENTIONS:
Behavioral: Cognitive functional therapy via tele rehabilitation — Participants in the CFT group will be treated by a physiotherapist with seventeen years of clinical experience and that has attended six CFT workshops with three of the international tutors of the method. She has completed 212 hours of training including workshops, patient examinations and a pilot study under the supervision of a physiotherapist with more than seven years of clinical experience in CFT. Another two physiotherapists, one with more than fifteen years and the other with more than ten years of clinical experience, and both with more than 106 hours of CFT training including CFT via tele physiotherapy, will complete the staff.
  Arms: Cognitive functional therapy (CFT) via tele rehabilitation
Other: Pilates via tele rehabilitation — Physiotherapist will have the freedom to judge about the exercises´ progression and the need of adaptation considering both the level of difficulty to perform each exercise according to the original proposal and the individual´s demands. The treating physiotherapists will have at least 2 years of clinical practice in Pilates and clinical experience in Pilates via teleconference.
  Arms: Pilates

SUMMARY:
There is evidence of three randomized controlled trials that face-to-face CFT reduces disability compared with active interventions for adults with chronic low back pain. The pandemic enabled the popularization of tele rehabilitation around the globe, but there are still no clinical trial testing the effectiveness of Cognitive Functional Therapy (CFT) via tele rehabilitation for elderly people with chronic low back pain. The aim of this study is to investigate the effectiveness of CFT compared with Pilates, both via tele rehabilitation in elderly patients with chronic low back pain.

DETAILED DESCRIPTION:
This will be a parallel-group randomized controlled trial with intention to treat analysis conducted via tele rehabilitation in Brazil. Two hundreds elderly people with chronic low back pain (except low risk on STartback screening tool) will be randomized to receive CFT (2 individualized sessions and 4-8 group sessions) or group Pilates (6-10 sessions) up to 12 weeks treatment. Participants will be assessed at baseline, post-intervention (12 weeks) 24 and 48 weeks after randomization. The trial will include cost-effectiveness and cost-utility analyses. Data of quality of life, healthcare costs, patient and family costs, and absenteism costs will be collected. The cost-effectiveness analysis will be performed using disability and pain intensity as outcomes. Costs and quality-adjusted life years will be used to calculate cost-utility.

Three qualitative studies will be conducted during the trial. The first will be performed by means of the interviews with a subsample of the participants before randomization. The aim will be to investigate how elderly people with chronic low back pain perceive their condition. The second will be performed by means of the analysis of a subsample of video recordings of CFT treatments. The aim will be to investigate the narratives of elderly people with chronic low back pain during CFT treatment sessions. The third will be performed after the last follow up by means of an interview with a subsample of participants that received CFT treatment. The aim will be to investigate the perceptions of elderly people with chronic low back pain about the impact of CFT via telerehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* A main complaint of pain in the area between the 12th rib and buttock crease with or without accompanying non-radicular leg pain;
* Episode of ongoing low back pain for at least 12 weeks' duration;
* Presenting to a primary care clinician at least 6 weeks ago for this episode of LBP;
* Being able to walk independently (with or without aids);
* Ability to understand Portuguese well enough to be able to fill in the questionnaires.
* Medium or high risk score on STartback screening tool.

Exclusion Criteria:

* Known or suspected red flag disorders like fracture, malignancy/cancer, cauda equina syndrome or progressive neurological disorder, inflammatory or infective diseases of the spine;
* Suspected radicular pain (dominant leg pain, positive neural tissue provocation tests and/or any two of altered strength, reflexes or sensation for the same nerve root, assessed clinically);
* Spinal surgery < 6 months previously;
* Invasive procedures for pain relief (ex: epidural injection, rhizotomy) in the last three months;
* Scoliosis (if considered the primary cause of pain);
* Unstable heart conditions;
* Chikungunya or Dengue virus disease transmitted by mosquitoes;
* Relevant cognition deficit measured by 10 point cognitive screener, with a cut-off point of less than 8 points, 18 for participants with elementary education, and 26 for participants with secondary and/or higher education;
* Post Covid-19 sequelae of pain.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-09-02 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Disability | 12 weeks after randomization
  Quebec Back Pain Disability Scale (0-100), higher scores mean worse outcome

SECONDARY OUTCOMES:
Pain intensity | 12 weeks, 24 weeks and 48 weeks after randomization
  Numerical Pain Rating Scale (0-10), higher scores mean a worse outcome
Disability | 24 weeks and 48 weeks after randomization
  Quebec Back Pain Disability Scale (0-100), higher scores mean a worse outcome
Function | 12 weeks, 24 weeks and 48 weeks after randomization
  Patient Specific Functional Scale (0-10), higher scores mean better outcome
Anxiety | 12 weeks, 24 weeks and 48 weeks after randomization
  Brief Psychosocial Questions (0-10), higher scores mean a worse outcome
Depression | 12 weeks, 24 weeks and 48 weeks after randomization
  Brief Psychosocial Questions (0-10),higher scores mean a worse outcome
Catastrophization | 12 weeks, 24 weeks and 48 weeks after randomization
  Brief Psychosocial Questions (0-10), higher scores mean a worse outcome
Fear of movement | 12 weeks, 24 weeks and 48 weeks after randomization
  Brief Psychosocial Questions (0-10), higher scores mean a worse outcome
Social isolation | 12 weeks, 24 weeks and 48 weeks after randomization
  Brief Psychosocial Questions (0-10), higher scores mean a worse outcome
Stress | 12 weeks, 24 weeks and 48 weeks after randomization
  Brief Psychosocial Questions (0-10), higher scores mean a worse outcome
Sleep disturbance | 12 weeks, 24 weeks and 48 weeks after randomization
  Subjective Health Complaints Inventory (0-3), higher scores mean a worse outcome
Costs | 12 weeks, 24 weeks and 48 weeks after randomization
  Assessments of healthcare costs, patients and family costs, and absenteeism costs by a specific questionnaire (total costs in £)
Quality-adjusted life years | 12 weeks, 24 weeks and 48 weeks after randomization
  SF-6D questionnaire (0-1), higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ney Meziat-Filho, PhD, Study Director — Centro Universitario Augusto Motta - UNISUAM
Locations (1):
- Centro Universitário Augusto Motta, Rio de Janeiro, Brazil

REFERENCES:
- [Background] O'Keeffe M, O'Sullivan P, Purtill H, Bargary N, O'Sullivan K. Cognitive functional therapy compared with a group-based exercise and education intervention for chronic low back pain: a multicentre randomised controlled trial (RCT). Br J Sports Med. 2020 Jul;54(13):782-789. doi: 10.1136/bjsports-2019-100780. Epub 2019 Oct 19. PMID 31630089
- [Background] Castro J, Correia L, Donato BS, Arruda B, Agulhari F, Pellegrini MJ, Belache FTC, de Souza CP, Fernandez J, Nogueira LAC, Reis FJJ, Ferreira AS, Meziat-Filho N. Cognitive functional therapy compared with core exercise and manual therapy in patients with chronic low back pain: randomised controlled trial. Pain. 2022 Dec 1;163(12):2430-2437. doi: 10.1097/j.pain.0000000000002644. Epub 2022 Apr 4. PMID 35384931
- [Background] Belache FTC, Souza CP, Fernandez J, Castro J, Ferreira PDS, Rosa ERS, Araujo NCG, Reis FJJ, Almeida RS, Nogueira LAC, Correia LCL, Meziat-Filho N. Trial Protocol: Cognitive functional therapy compared with combined manual therapy and motor control exercise for people with non-specific chronic low back pain: protocol for a randomised, controlled trial. J Physiother. 2018 Jul;64(3):192. doi: 10.1016/j.jphys.2018.02.018. Epub 2018 Jun 11. PMID 29903598
- [Background] Caneiro JP, Smith A, Bunzli S, Linton S, Moseley GL, O'Sullivan P. From Fear to Safety: A Roadmap to Recovery From Musculoskeletal Pain. Phys Ther. 2022 Feb 1;102(2):pzab271. doi: 10.1093/ptj/pzab271. PMID 34971393
- [Background] Fernandez J, Ferreira AS, Castro J, Correia LCL, Meziat-Filho N. Comment on the paper "Cognitive functional therapy in patients with non specific chronic low back pain", by Vibe Fersum et al. Eur J Pain. 2019 Sep;23(8):1574-1575. doi: 10.1002/ejp.1441. Epub 2019 Jun 26. No abstract available. PMID 31190411
- [Background] Miki T, Kondo Y, Kurakata H, Buzasi E, Takebayashi T, Takasaki H. The effect of cognitive functional therapy for chronic nonspecific low back pain: a systematic review and meta-analysis. Biopsychosoc Med. 2022 May 21;16(1):12. doi: 10.1186/s13030-022-00241-6. PMID 35597961
- [Background] Vibe Fersum K, O'Sullivan P, Skouen JS, Smith A, Kvale A. Efficacy of classification-based cognitive functional therapy in patients with non-specific chronic low back pain: a randomized controlled trial. Eur J Pain. 2013 Jul;17(6):916-28. doi: 10.1002/j.1532-2149.2012.00252.x. Epub 2012 Dec 4. PMID 23208945
- [Background] American College of Sports Medicine Position Stand. Exercise and physical activity for older adults. Med Sci Sports Exerc. 1998 Jun;30(6):992-1008. PMID 9624662
- [Background] Kent P, Mirkhil S, Keating J, Buchbinder R, Manniche C, Albert HB. The concurrent validity of brief screening questions for anxiety, depression, social isolation, catastrophization, and fear of movement in people with low back pain. Clin J Pain. 2014 Jun;30(6):479-89. doi: 10.1097/AJP.0000000000000010. PMID 24281277
- [Background] GBD 2016 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 328 diseases and injuries for 195 countries, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2017 Sep 16;390(10100):1211-1259. doi: 10.1016/S0140-6736(17)32154-2. PMID 28919117
- [Background] Fernandez J, Lunkes LC, Meziat-Filho N. Biopsychosocial approaches to telerehabilitation for chronic primary musculoskeletal pain: A real possibility for physical therapists, that is here to stay. Braz J Phys Ther. 2022 Jan-Feb;26(1):100350. doi: 10.1016/j.bjpt.2021.04.011. Epub 2021 May 9. No abstract available. PMID 34001421